CLINICAL TRIAL: NCT03180359
Title: Vaccines Immunogenicity in Children Transplanted or Candidate for a Renal, Hepatic, Cardiac or Pulmonary Transplantation, Followed in the Rhône-Alpes Region. A Descriptive and Prospective Monocentric Cohort Study
Brief Title: Vaccines Immunogenicity in Renal, Hepatic, Cardiac or Pulmonary Transplanted Children
Acronym: COVAGREF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0354; 2015-A00854-45 (Other: ID-RCB)
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Transplantation
Keywords: solid transplant; grafted children; vaccine recommendation; immunization efficacy; solid grafted children; solid transplant candidate children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient already transplanted or waiting for a transplantation (Experimental)
  Interventions: Biological: Recommended vaccine scheme according to French Vaccine Schedule 2015

INTERVENTIONS:
Biological: Recommended vaccine scheme according to French Vaccine Schedule 2015 — * BCG
  * Measles mumps rubella (MMR)
  * Varicella (chicken pox)
  * Rotavirus
  * Seasonal flu (live vaccine delivered nasally and inactivated vaccine injectable)
  * Yellow Fever
  * Diphteria tetanus poliomyelitis whopping cough (DTwP)
  * Haemophilus influenzae type b
  * Hepatitis B
  * Meningococcus conjugate
  * Pneumococcus
  * Human papillomavirus
  * Hepatitis A
  Vaccine administration would be done according to French Vaccine Schedule 2015 for mainstream population and for grafted children or transplant candidate children

SUMMARY:
Thanks to improved surgical techniques, postoperative management and immunosuppressive therapies, an increasing number of children benefit from renal, hepatic, cardiac and pulmonary transplantation. Infection is a significant cause of mortality and morbidity in these patients, particularly due to vaccine-preventable diseases. Vaccination is one of the effective means of reducing infection-related mortality in these particularly vulnerable children. It is mostly well-tolerated, but all the more effective as it is performed early before transplantation, at best during a dedicated consultation, according to a vaccine scheme adapted to the immunocompromised child. In the almost constant absence of clinical efficacy data in populations of immunocompromised individuals, vaccine efficacy is most often indirectly estimated by immunogenicity, using protective correlates obtained by extrapolation in immunocompetent individuals.

Primary objective: To estimate the immunogenicity of vaccines recommended in children transplanted or candidate for renal, hepatic, cardiac and pulmonary transplantation, using serological titers measurements before and after a vaccine injection for: influenza, pneumococcus, chicken pox, measles, tetanus, hepatitis A and hepatitis B.

These serological titers will be compared to correlates of protection existing for each valency.

The evolution of serological titers will be described during the first year. The vaccination will be carried out within the routine care, according to the recommendations.

Secondary objectives:

* describe and quantify the vaccination status of patients
* describe the vaccination coverage of their entourage
* evaluate the tolerance and efficacy of vaccines

ELIGIBILITY:
Inclusion Criteria:

* children and adolescent between 0 and 17 years old
* registered in the database of the Agency of Biomedicine
* transplanted or waiting for a renal, hepatic, cardiac or pulmonary transplantation
* followed up in the Rhône-Alpes region between January 1st , 2015 and December 31th, 2016
* patients requiring vaccination in standard care

Exclusion Criteria:

* adults
* children or adolescent not able not comply with protocol
* children, adolescent or patient parents or legal guardian not opposed to study participation

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-10-13 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of vaccines recommended in children transplanted or candidate for renal, hepatic, cardiac and pulmonary transplantation | at Month 0
  The immunogenicity is appraised from serological titer before and after vaccine injection. These serological titers will be compared to existing reference protection correlates for each valency, and defined as protective or non-protective: Tetanus (>0,1 UI/ml), hepatitis B (>10 mUI/ml), hepatitis A (> 20 mUI/ml), measles (0,18 in EIA index), chicken pox (> 5 gp Elisa UI/ml or > 50 UI/l with an highly sensitive test), influenza (Hemagglutination Inhibition Assay > 1/40), pneumococcus (0,35 µg/ml, > 0,4 mg/l for each specific serotype, if > 2/3 or 4/6, protecting serotype)
Immunogenicity of vaccines recommended in children transplanted or candidate for renal, hepatic, cardiac and pulmonary transplantation | between Month 1 and Month 3
  The immunogenicity is appraised from serological titer before and after vaccine injection. These serological titers will be compared to existing reference protection correlates for each valency, and defined as protective or non-protective: Tetanus (>0,1 UI/ml), hepatitis B (>10 mUI/ml), hepatitis A (> 20 mUI/ml), measles (0,18 in EIA index), chicken pox (> 5 gp Elisa UI/ml or > 50 UI/l with an highly sensitive test), influenza (Hemagglutination Inhibition Assay > 1/40), pneumococcus (0,35 µg/ml, > 0,4 mg/l for each specific serotype, if > 2/3 or 4/6, protecting serotype)
Immunogenicity of vaccines recommended in children transplanted or candidate for renal, hepatic, cardiac and pulmonary transplantation | Month 12
  The immunogenicity is appraised from serological titer before and after vaccine injection. These serological titers will be compared to existing reference protection correlates for each valency, and defined as protective or non-protective: Tetanus (>0,1 UI/ml), hepatitis B (>10 mUI/ml), hepatitis A (> 20 mUI/ml), measles (0,18 in EIA index), chicken pox (> 5 gp Elisa UI/ml or > 50 UI/l with an highly sensitive test), influenza (Hemagglutination Inhibition Assay > 1/40), pneumococcus (0,35 µg/ml, > 0,4 mg/l for each specific serotype, if > 2/3 or 4/6, protecting serotype)
Immunogenicity of vaccines recommended in children transplanted or candidate for renal, hepatic, cardiac and pulmonary transplantation | 3-month post-transplantation (if transplantation occurs during the study)
  The immunogenicity is appraised from serological titer before and after vaccine injection. These serological titers will be compared to existing reference protection correlates for each valency, and defined as protective or non-protective: Tetanus (>0,1 UI/ml), hepatitis B (>10 mUI/ml), hepatitis A (> 20 mUI/ml), measles (0,18 in EIA index), chicken pox (> 5 gp Elisa UI/ml or > 50 UI/l with an highly sensitive test), influenza (Hemagglutination Inhibition Assay > 1/40), pneumococcus (0,35 µg/ml, > 0,4 mg/l for each specific serotype, if > 2/3 or 4/6, protecting serotype)

SECONDARY OUTCOMES:
Levels of blood antibodies corresponding to the following vaccine valencies: influenza, pneumococcus, chicken pox (varicella), measles, tetanus, hepatitis A and hepatitis B. | at Month 0
Levels of blood antibodies corresponding to the following vaccine valencies: influenza, pneumococcus, chicken pox (varicella), measles, tetanus, hepatitis A and hepatitis B. | between Month 1 and Month 3
Levels of blood antibodies corresponding to the following vaccine valencies: influenza, pneumococcus, chicken pox (varicella), measles, tetanus, hepatitis A and hepatitis B. | at Month 12
Levels of blood antibodies corresponding to the following vaccine valencies: influenza, pneumococcus, chicken pox (varicella), measles, tetanus, hepatitis A and hepatitis B. | 3-month post-transplantation (if transplantation occurs during the study)
the number of early or late injections | at Month 0,
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of missing injections and supplementary injections | at Month 0,
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of days in advance or delayed from recommended injections (per injection and cumulative) | at Month 0,
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of early or late injections | between Month 1 and Month 3
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of missing injections and supplementary injections | between Month 1 and Month 3
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of days in advance or delayed from recommended injections (per injection and cumulative) | between Month 1 and Month 3
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of early or late injections | at Month 12
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of missing injections and supplementary injections | at Month 12
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
the number of days in advance or delayed from recommended injections (per injection and cumulative) | at Month 12
  Vaccine status compliance with vaccine recommendation, from literature data and from the opinion of the Vaccine Technical Committee President.
  Compliance will be appraised by considering for each valence:
  * the number of early or late injections
  * the number of missing injections and supplementary injections
  * the number of days in advance or delayed from recommended injections (per injection and cumulative) 2 age groups will be differentiate : <2 years (primary vaccination) and >2 years For each age group, early or late injections are defined by considering literature data and the opinion of the Vaccine Technical Committee President.
Vaccination coverage of patients' entourage | at month 0
  Number of missing, additional, early or late injections, compared to vaccine recommendations.
Patients' vaccine tolerance | at Week 1
  Local reactions, fever, clinical or biological signs of rejection
Patients' vaccine tolerance | at Month 1 after injection
  Local reactions, fever, clinical or biological signs of rejection

CONTACTS AND LOCATIONS:
Overall Officials: Laure HEES, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No